CLINICAL TRIAL: NCT03338582
Title: STIMulation Cardiaque et TAVI : évolution Des Troubles Conductifs Atrio-ventriculaires après TAVI
Brief Title: STIMTAVI : Evolution of Atrioventricular Conduction Disorders After TAVI
Acronym: STIMTAVI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Association de Recherche en Cardiologie des Alpes (Other)
Collaborators: LivaNova (Industry)
Responsible Party: Sponsor
Other Study IDs: ARCAlpes
Record Dates: First submitted 2017-10-20; First posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Pacemaker Implantation; TAVI
Keywords: Pacemaker; Conduction disturbance; TAVI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators propose to carry out an observational study of patients implanted with a pacemaker using AAI SafeR® mode after a TAVI procedure. This study aims to define the persistence or not of high-grade AVB beyond seven days after the procedure, based on the analysis of PM memories, and define definitive cardiac pacing indications after TAVI procedure.

DETAILED DESCRIPTION:
Atrioventricular (A-V) conduction disorders are common after Transcatheter Aortic Valve Implantation (TAVI) and the average of a pacemaker implantation after TAVI is 15% to 17%.

The European Society of Cardiology recommends to implant a permanent pacemaker (PM) in case of persistant high-grade A-V block (AVB) within 7 days of a TAVI procedure (class I recommendation, level of evidence C).

Some conduction disturbances are transient and might not need a definitive indication for pacemaker implantation. A recent study, based on dependency of patients to pacing, estimate that in half the patients, conduction disturbances that led to the implantation of a pacemaker after TAVI procedure would have disappear 30 days after the procedure.

Many studies tried to better define the indications of these devices. However, their evaluation criteria do not allow to prove these pacemakers were useful, because these studies are mainly based on the rate of implantation of pacemakers, or on the percentage of ventricular pacing. These studies may overestimate the usefulness of the pacemaker because of unnecessary ventricular pacing, or underestimate it in patients with high grade paroxysmal AVB, that could have been responsible for syncope or death.

Today some pacemakers allow a better occurrence of spontaneous A-V conduction and monitor precisely the atrioventricular conduction.

The AAI SafeR® mode from Sorin® allows the pacemaker to switch from a single to a dual chamber mode in case of AVB; these switches are stored in the memories of PM as endocardial electrogram (EGM) which can be validated afterwards. The use of this algorithm could allow an accurate assessment of the persistence of high level conduction disturbances in patients implanted with a pacemaker after a TAVI procedure. A study published in late 2014 using this tool in monitoring post TAVI conduction disorders on a small number of patients, other studies used the same tool in other cardiac pathologies.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years who underwent implantation of a TAVI and that were implanted during the hospitalization with a dual chamber pacemaker Sorin®, set in AAI SafeR ® or AAI SafeR-R® mode.

Exclusion Criteria:

* Patients with life expectancy at hospital discharge estimated as less than 1 year
* TAVI procedure failure
* Patients refusing to be involved in the study
* Patients implanted with a PM of a brand different than Sorin® during the hospital phase or implanted Sorin® PM but not set in a AAI or AAI SafeR SafeR-R mode
* Patients with PM implant before TAVI
* Permanent AF at the implantation time
* Patients with Single or Triple chamber PM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 275 patients over 18 years who underwent implantation of a TAVI and that were implanted during the hospitalization with a dual chamber pacemaker Sorin®, set in AAI SafeR ® or AAI SafeR-R® mode.
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2018-01-19 (Estimated); Study Completion 2018-04-19 (Estimated)

PRIMARY OUTCOMES:
To look for one or several high level A-V block episodes beyond seven days after a TAVI procedure, by the analysis of the EKG and of the pacemaker memories during the follow-up visits | Until the completion of the study (first follow-up visit 1 to 3 months after TAVI, last follow-up visit 1 year after TAVI)
  High level A-V Block in patients after TAVI procedure is defined:
  * Either by the analysis of the pacemaker memories during the follow-up visits showing the switches from AAI Safe-R to DDD mode after one or more of these three reasons:
    * a succession of at least 2 consecutive blocked P waves
    * more than 3 blocked P waves among 12 consecutive cycles
    * ventricular pause for over 2 seconds with at least one blocked P wave
  * Either by the presence of a high level AVB on the EKG during the follow-up visit (pacemaker temporally set to DDI 30 bpm mode)
  We classify as transitional AVB (D7 persistent, non-persistent beyond 1 month), and permanent AVB (persistent beyond 1 month).

SECONDARY OUTCOMES:
To study the influence of certain predefined factors on the risk of high-level A-V block after a TAVI procedure. | An average of 8 days (from the day before the TAVI procedure to 7 days after TAVI)
  In accordance with the secondary objective, we will study the influence of certain predefined factors on the risk of high-level A-V block after a TAVI procedure : preexisting conduction disturbances (complete right bundle branch block, left anterior hemiblock, first degree A-V block), high grade AVB during the TAVI procedure, worsening of conduction disturbances during the procedure or within the next hour (appearance of a left bundle branch block, QRS widening beyond 120ms, prolongation of PR beyond 200ms ), lengthening of the HV interval immediately after the procedure TAVI or later (if an electrophysiological study is performed), implantation of a Medtronic® CoreValve prosthesis (compared to an Edwards® Sapien prosthesis), height of the implantation of the valve, oversizing.

CONTACTS AND LOCATIONS:
Overall Officials: Didier IRLES, Dr, Study Director — Association de Recherche en Cardiologie des Alpes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Irles D, Salerno F, Cassagneau R, Eschalier R, Maupain C, Dupuis JM, Mansourati J, Guedon L, Marijon E, Frey P; Other members of the STIMulation cardiaque post-TAVI (STIM-TAVI) study. Evolution of high-grade atrioventricular conduction disorders after transcatheter aortic valve implantation in patients who underwent implantation of a pacemaker with specific mode-that minimizes ventricular pacing-activated. J Cardiovasc Electrophysiol. 2021 May;32(5):1376-1384. doi: 10.1111/jce.14970. Epub 2021 Mar 4. PMID 33625762

DOCUMENTS (1):
  • Study Protocol (2015-10-15): https://cdn.clinicaltrials.gov/large-docs/82/NCT03338582/Prot_000.pdf